CLINICAL TRIAL: NCT03167333
Title: Does Synovitis Affect Treatment Efficacy in Intra-articular Injection Therapy to Osteoarthritis
Brief Title: The Role of Synovitis in Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-03-009B
Record Dates: First submitted 2017-05-18; First posted 2017-05-25 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Synovitis of Knee; Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP group (Experimental): the patients received PRP(platelet-rich-plasma) injection twice at 2-week intervals
  Interventions: Drug: platelet rich plasma
- HA group (Active Comparator): the patients received HA(hyaluronic acid) injection twice at 2-week intervals
  Interventions: Drug: Hyaluronic acid

INTERVENTIONS:
Drug: platelet rich plasma — The amount of PPR was about 4-5 cc
  Arms: PRP group
Drug: Hyaluronic acid — HA was 2.5cc
  Arms: HA group

SUMMARY:
To determine whether platelet-rich-plasma (PRP) or HA (hyaluronic acid)injection into synovitis in osteoarthritis(OA) knee can achieve improvement in knee function and reduce synovitis.

DETAILED DESCRIPTION:
Methods:

sixty patients with OA knee having unilateral or bilateral synovitis validated by ultrasound (N=40) were studied. All the patients were randomized to receive PRP (N=40) or Hyaluronic acid(HA)(N=40) injection twice at 2-week intervals; Clinical assessments were performed using a visual analog scale(VAS) and The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC index) before injection at baseline, 4 weeks(first evaluation) and 12 weeks(secondary evaluation). Imaging evaluation based on color Doppler ultrasound(CDUS) and the depth of synovial fluid accumulation ,and the width of synovial hypertrophy was performed simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with OA knee according to ACR guideline

  1. stiffness less than 30min
  2. cracking sound during activity
  3. more than 30min pain for last 2 months
  4. non-bed ridden patients
  5. no structure abnormality
  6. synovitis was proved by US

Exclusion Criteria:

1. OA knee secondary to other disease 2 . more than 10 years after diagnosing OA 3. under knee surgery within 3 months 4. autoimmune disease 5. refuses inform/consent process

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
visual analog scale(VAS) | before injection at baseline
visual analog scale(VAS) | 4 weeks(first evaluation)
visual analog scale(VAS) | 12 weeks(secondary evaluation)
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC index) | before injection at baseline
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC index) | 4 weeks(first evaluation)
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC index) | 12 weeks(secondary evaluation)

SECONDARY OUTCOMES:
Imaging evaluation based on color Doppler ultrasound(CDUS) and the depth of synovial fluid accumulation ,and the width of synovial hypertrophy was performed simultaneously. | before injection at baseline
Imaging evaluation based on color Doppler ultrasound(CDUS) and the depth of synovial fluid accumulation ,and the width of synovial hypertrophy was performed | 4 weeks(first evaluation)
Imaging evaluation based on color Doppler ultrasound(CDUS) and the depth of synovial fluid accumulation ,and the width of synovial hypertrophy was performed | 12 weeks(secondary evaluation)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei veteran general hospital yuli branch, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided